CLINICAL TRIAL: NCT00282152
Title: Safety and Tolerability of Neurostimulation in Early Stage Parkinson's Disease
Brief Title: Deep Brain Stimulation (DBS) for Early Stage Parkinson's Disease (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Charles, Associate Professor of Neurology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 040797; 1363 (Other: Clinical Research Center); G050016 (Other: FDA IDE)
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
Keywords: Early Stage Parkinson's Disease; Parkinson's Disease; Deep Brain Stimulation; PD; DBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ODT (Active Comparator): Optimal drug therapy: The drugs used on this study are not investigational. They are drugs for Parkinson's disease that are standard of care. The drug form, dosage, frequency and duration will vary.
  Interventions: Drug: Optimal drug therapy
- DBS+ODT (Experimental): Subjects receive bilateral subthalamic nucleus (B-STN) DBS and continue to take optimal drug therapy as prescribed by their treating neurologist.
  B-STN DBS: Deep brain stimulation (DBS) of both the right and left sub-thalamic nucleus (STN) is an FDA approved treatment for mid- and advanced PD. DBS is not approved for early stage PD. In mid- and advanced stage Parkinson's disease, using DBS in this area of the brain lessens symptoms and allows patients to take less drug to control the disease. Dosage and frequency are not applicable to the DBS. Once the DBS is placed, unless deemed necessary, it will not be removed.
  Optimal drug therapy: The drugs used on this study are not investigational. They are drugs for Parkinson's disease that are standard of care. The drug form, dosage, frequency and duration will vary.
  Interventions: Device: B-STN DBS; Drug: Optimal drug therapy

INTERVENTIONS:
Device: B-STN DBS — Deep brain stimulation (DBS) of both the right and left sub-thalamic nucleus (STN) is an FDA approved treatment for advanced PD. In mid- and advanced stage Parkinson's disease, using DBS in this area of the brain lessens symptoms and allows patients to take less drug to control the disease. Dosage and frequency are not applicable to the DBS. Once the DBS is placed, unless deemed necessary, it will not be removed.
  Arms: DBS+ODT
Drug: Optimal drug therapy — The drugs used on this study are not investigational. They are drugs for Parkinson's disease that are standard of care. The drug form, dosage, frequency and duration will vary. Examples of drugs used include carbidopa/levodopa, pramipexole, ropinirole, and selegiline.

SUMMARY:
Bilateral subthalamic nucleus deep brain stimulation (B-STN DBS) is one of the most effective surgical treatments for PD patients suffering from levodopa-induced motor complications. The relatively low incidence of permanent adverse effects and the potential for neuroprotection and alteration of the natural course of PD suggest a highly favorable benefit-to-risk ratio of this procedure. Since neuroprotection is best applied early in the disease course when there are more surviving neurons, we believe that further investigation of this procedure is warranted. The proposed pilot study will provide the necessary data to substantiate the safety and tolerability of the procedure as well as provide data for the design of a full-scale, multicenter trial to investigate the hypothesis that B-STN DBS is a safe and effective treatment to slow the progression of PD.

DETAILED DESCRIPTION:
This pilot trial is designed specifically to collect the preliminary safety and tolerability data necessary to conduct a future phase III clinical trial to investigate the hypothesis that deep brain stimulation of the subthalamic nucleus in subjects with early Parkinson's will slow the progression of the disease.

The study design is a prospective, randomized, blinded, single-center trial comparing the safety and tolerability of B-STN DBS + Optimal Drug Therapy (ODT) vs. (ODT) alone (control, standard of care) in 30 subjects (15 per group) with early PD (Hoehn and Yahr stage II when off medication).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of probable idiopathic PD.
* Demonstrated response to dopaminergic therapy, defined as demonstrating at least 30% improvement in parkinsonian motor signs, based upon the UPDRS motor examination subscore, following the administration of their dopamine agonist (DA) drug(s) during the screening neurological examination.
* Hoehn and Yahr (H&Y) stage II when OFF medication.
* No contraindications to surgery.
* Age between 50 and 75 years old.
* Available for follow-up for four years.
* Informed Consent: The subject understands the risks, benefits, and alternatives to the study procedures and participation in the study.
* MRI within normal range for age.
* Levodopa or dopamine agonist therapy for greater than six months but less than or equal to four years.

Exclusion Criteria:

* Evidence of an alternative diagnosis or secondary parkinsonism, as suggested by features unusual early in the clinical course: Prominent postural instability, freezing phenomena, or hallucinations unrelated to medications in the first 3 years after symptom onset; dementia preceding motor symptoms; supranuclear gaze palsy (other than restriction of upward gaze) or slowing of vertical saccades in the first year; severe, symptomatic dysautonomia unrelated to medications; documentation of a condition known to produce parkinsonism and plausibly connected to the subject's symptoms (such as suitably located focal brain lesions or neuroleptic use within the past 6 months)
* Uncontrolled medical condition or clinically significant medical disease that would increase the risk of developing pre- or postoperative complications (e.g., significant cardiac or pulmonary disease, uncontrolled hypertension).
* Evidence of dementia
* Major psychiatric disorder
* Previous brain operation or injury.
* Active participation in another clinical trial for the treatment of PD.
* Patients who have demand cardiac pacemakers or implantable cardioverter defibrillators (ICD's).
* Patients who have medical conditions that require repeat MRI scans or diathermy treatments.
* Evidence of existing dyskinesias or motor fluctuations.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-03; Primary Completion 2012-01 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. David Charles, MD, Principal Investigator — Vanderbilt University Department of Neurology

REFERENCES:
- [Derived] Hacker ML, Meystedt JC, Turchan M, Cannard KR, Harper K, Fan R, Ye F, Davis TL, Konrad PE, Charles D. Eleven-Year Outcomes of Deep Brain Stimulation in Early-Stage Parkinson Disease. Neuromodulation. 2023 Feb;26(2):451-458. doi: 10.1016/j.neurom.2022.10.051. Epub 2022 Dec 24. PMID 36567243
- [Derived] Hacker ML, Turchan M, Heusinkveld LE, Currie AD, Millan SH, Molinari AL, Konrad PE, Davis TL, Phibbs FT, Hedera P, Cannard KR, Wang L, Charles D. Deep brain stimulation in early-stage Parkinson disease: Five-year outcomes. Neurology. 2020 Jul 28;95(4):e393-e401. doi: 10.1212/WNL.0000000000009946. Epub 2020 Jun 29. PMID 32601120
- [Derived] Millan SH, Hacker ML, Turchan M, Molinari AL, Currie AD, Charles D. Subthalamic Nucleus Deep Brain Stimulation in Early Stage Parkinson's Disease Is Not Associated with Increased Body Mass Index. Parkinsons Dis. 2017;2017:7163801. doi: 10.1155/2017/7163801. Epub 2017 Jun 6. PMID 28676842
- [Derived] Charles PD, Dolhun RM, Gill CE, Davis TL, Bliton MJ, Tramontana MG, Salomon RM, Wang L, Hedera P, Phibbs FT, Neimat JS, Konrad PE. Deep brain stimulation in early Parkinson's disease: enrollment experience from a pilot trial. Parkinsonism Relat Disord. 2012 Mar;18(3):268-73. doi: 10.1016/j.parkreldis.2011.11.001. Epub 2011 Nov 21. PMID 22104012

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants excluded prior to treatment ( 1 withdrew consent and 6 failed screening)
Groups:
- Optimal Drug Therapy (ODT): Patients receive optimal drug therapy as prescribed by their treating neurologist.
  Optimal drug therapy: The drugs used on this study are not investigational. They are drugs for Parkinson's disease that are standard of care. The drug form, dosage, frequency and duration will vary. Examples of drugs used include carbidopa/levodopa, pramipexole, ropinirole, and selegiline.
- Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT): Subjects receive bilateral subthalamic nucleus (B-STN) DBS and continue to take optimal drug therapy as prescribed by their treating neurologist.
  B-STN DBS: Deep brain stimulation (DBS) of both the right and left sub-thalamic nucleus (STN) is an FDA approved treatment for mid- and advanced PD. DBS is not approved for early stage PD. In mid- and advanced stage Parkinson's disease, using DBS in this area of the brain lessens symptoms and allows patients to take less drug to control the disease. Dosage and frequency are not applicable to the DBS. Once the DBS is placed, unless deemed necessary, it will not be removed.
  Optimal drug therapy: The drugs used on this study are not investigational. They are drugs for Parkinson's disease that are standard of care. The drug form, dosage, frequency and duration will vary. Examples of drugs
Period: Overall Study
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Full Range); unit: years] | 60 [51 to 69] | 60 [52 to 74] | 60 [51 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 13 | 14 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Safety: Time to Reach a 4 Point Increase (Worsening) in Unified Parkinson's Disease Rating Scale (UPDRS) Motor Score
Description: The primary hypothesis of this feasibility trial was focused on safety and tolerability and that the DBS+ODT group would not worsen more quickly than the ODT group.
Time Frame: baseline to 24 months
Population: all 29 subjects that completed at least one follow up visit were included in the primary analysis following intent to treat principle
Measure: Mean (95% Confidence Interval); unit: months
Groups:
- Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT): Subjects receive bilateral subthalamic nucleus (B-STN) DBS and continue to take optimal drug therapy as prescribed by their treating neurologist.
  B-STN DBS: Deep brain stimulation (DBS) of both the right and left sub-thalamic nucleus (STN) is an FDA approved treatment for mid- and advanced PD. DBS is not approved for early stage PD. In mid- and advanced stage Parkinson's disease, using DBS in this area of the brain lessens symptoms and allows patients to take less drug to control the disease. Dosage and frequency are not applicable to the DBS. Once the DBS is placed, unless deemed necessary, it will not be removed.
  Optimal drug therapy: The drugs used on this study are not investigational. They are drugs for Parkinson's disease that are standard of care. The drug form, dosage, frequency and duration will vary.
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
Number analyzed (Participants) | 14 | 15
months | 15 [10.7 to 19.3] | 14.1 [10.3 to 18]
Statistical Analysis 1: Comparison: Optimal Drug Therapy (ODT) vs Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT); Test type: Non-Inferiority — Because the purpose of this trial was to provide preliminary safety and tolerability data, the primary hypothesis was that the DBS+ODT group would not worsen more quickly than the ODT group. The primary endpoint was defined as the time to reach a four-point worsening of the UPDRS-III score following a one week treatment washout as assessed by the blinded rater; p = 0.968, Log Rank

2. Primary Outcome: Levodopa Equivalents, Change From Baseline
Description: 100 mg of levodopa with a dopa-decarboxylase inhibitor = 133 mg of controlled-release levodopa preparations = total levodopa dose + (total levodopa dose x 0.33) of levodopa with dopa-decarboxylase and entacapone = 1 mg of pergolide, pramipexole, or lisuride = 5 mg of ropinirole = 3.3 mg of rotigotine
Time Frame: baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: mg
Groups:
- Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT): Subjects receive B-STN DBS and continue to take optimal drug therapy as prescribed by their treating neurologist.
  B-STN DBS: Deep brain stimulation (DBS) of both the right and left sub-thalamic nucleus (STN) is an FDA approved treatment for advanced PD. DBS is not approved for early stage PD. The STN is a part of the brain that is very small in size and is located in the middle of the right and left sides of the brain. In this disease, this part of the brain becomes overactive and causes the symptoms of PD. It is thought that using DBS in this area of the brain lessens symptoms and allows patients to take less drug to control the disease. Dosage and frequency are not applicable to the DBS. Once the DBS is placed, unless deemed necessary, it will not be removed.
  Optimal drug therapy: The drugs used on this study are not investigational. They are drugs for Parkinson's disease that are standard of care. The drug form, dosage, frequency and duration will vary. Examples of drugs
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
Number analyzed (Participants) | 14 | 15
mg | 214.5 [16.9 to 412.1] | 97.7 [-93.7 to 288.7]
Statistical Analysis 1: Comparison: Optimal Drug Therapy (ODT) vs Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT); Study power was calculated based on the amount of PD medication consumed. We anticipated that the control group (ODT) would have a baseline value of 400 which would increase to 600, and that the treated group (DBS+ODT) would decrease from 400 to 300. A sample size of 12 patients per group (n=15, assuming 20% drop out) would have 80% power to detect a difference in means of 300 assuming that the common standard deviation is 250 using a two group t-test with a 0.05 two-sided significance level; Test type: Other; p = 0.40, t-test, 2 sided

3. Secondary Outcome: Change in UPDRS Part I, Mentation Behavior and Mood
Description: Score: 0-16 0 =normal, 16 = most disability
Time Frame: baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
Number analyzed (Participants) | 14 | 15
units on a scale | 1.1 [-0.1 to 2.3] | 1.2 [0.1 to 2.3]

4. Secondary Outcome: Change in UPDRS Part II, Activities of Daily Living
Description: Score: 0-52 0 =normal, 52 = most limited
Time Frame: baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
Number analyzed (Participants) | 14 | 15
units on a scale | 2.3 [-1.2 to 5.8] | 4.1 [0.7 to 7.5]

5. Secondary Outcome: Change in UPDRS Part III, Motor Examination, Excluding Rigidity
Description: Score: 0-56 0 = full movement, 56 = most limited
Time Frame: baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
Number analyzed (Participants) | 14 | 15
change in units on a scale | 3.4 [-2.9 to 9.8] | 0.1 [-6 to 6.1]

6. Secondary Outcome: Change in UPDRS Part IV, Complications of Therapy
Description: Score: 0-23 0 =no complications, 23 = most complications
Time Frame: baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
Number analyzed (Participants) | 14 | 15
units on a scale | 1.9 [0.4 to 3.4] | 0.3 [-1.2 to 1.7]

7. Secondary Outcome: Change in Total UPDRS
Description: The Total Unified Parkinson's Disease Rating Scale (UPDRS) is a composite scale, consisting of four sections that evaluate mood and behavior, activities of daily living, motor symptoms, and complications of medical therapy.
  Range is 0 to 16, with 16 being maximal disability
Time Frame: baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
Number analyzed (Participants) | 14 | 15
units on a scale | 8.4 [-0.3 to 17] | 5.63 [-2.6 to 13.9]

ADVERSE EVENTS:
Time Frame: baseline to 24 months
Arm/Group | Optimal Drug Therapy (ODT) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 2/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal Drug Therapy (ODT) (N=14) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT) (N=15)
Perioperative infarction in left basil ganglia (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) — Developed due to injury at subject's home.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Optimal Drug Therapy (ODT) (N=15) | Deep Brain Stimulation (DBS) Plus Optimal Drug Therapy (ODT) (N=15)
Insomnia (Nervous system disorders) | 5/14 (7) | 8 (8)
Nausea (Gastrointestinal disorders) | 6/14 (10) | 3 (3)
Nasopharyngitis (Immune system disorders) | 2/14 (3) | 5 (7)
Weight decreased (General disorders) | 6/14 (6) | 3 (3)
Dizziness (Nervous system disorders) | 5/14 (7) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3/14 (3) | 4 (5)
Weight increased (General disorders) | 5/14 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4/14 (4) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 3/14 (3) | 3 (3)
Fatigue (General disorders) | 2/14 (2) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 4/14 (4) | 1 (1)
Headache (Nervous system disorders) | 1/14 (2) | 1 (3)
Constipation (Gastrointestinal disorders) | 3/14 (3) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2/14 (2) | 2 (2)
Memory impairment (Nervous system disorders) | 1/14 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 2 (3)
Chest pain (Cardiac disorders) | 3/14 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3/14 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3/14 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2/14 (2) | 1 (1)
Hallucination (Nervous system disorders) | 2/14 (2) | 1 (1)
Pain in extremity (Nervous system disorders) | 2/14 (2) | 1 (1)
Somnolence (Nervous system disorders) | 2/14 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1/14 (1) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 2 (2)
Decreased appetite (General disorders) | 1/14 (1) | 2 (2)
Depression (Psychiatric disorders) | 0/14 (0) | 3 (3)
Abnormal touch sensation (Nervous system disorders) | 0/14 (0) | 3 (3)
Implant site pain (Surgical and medical procedures) | 0/14 (0) | 3 (3)
Aphasia (Nervous system disorders) | 2/14 (2) | 0 (0)
Diplopia (Eye disorders) | 2/14 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2/14 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2/14 (2) | 0 (0)
Hot flush (General disorders) | 2/14 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2/14 (2) | 0 (0)
Vision blurred (Nervous system disorders) | 2/14 (2) | 0 (0)
Oropharyngeal pain (Gastrointestinal disorders) | 1/14 (2) | 0 (0)
Agitation (Nervous system disorders) | 1/14 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/14 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1/14 (1) | 1 (1)
Incision site pain (Surgical and medical procedures) | 1/14 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1/14 (1) | 1 (1)
Pain (General disorders) | 1/14 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1/14 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0/14 (0) | 1 (2)
Confusional state (Nervous system disorders) | 0/14 (0) | 2 (2)
Influenza (Infections and infestations) | 0/14 (0) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 0/14 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/14 (0) | 2 (2)
Restlessness (General disorders) | 0/14 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0/14 (0) | 2 (2)
Abnormal dreams (Nervous system disorders) | 1/14 (1) | 0 (0)
Allergic rhinitis (Immune system disorders) | 1/14 (1) | 0 (0)
Asthenia (Nervous system disorders) | 1/14 (1) | 0 (0)
Blood pressure fluctuation (Cardiac disorders) | 1/14 (1) | 0 (0)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1/14 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1/14 (1) | 0 (0)
Dysphonia (General disorders) | 1/14 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1/14 (1) | 0 (0)
Gastric ulcers (Gastrointestinal disorders) | 1/14 (1) | 0 (0)
Gastrointestinal oedema (Gastrointestinal disorders) | 1/14 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1/14 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1/14 (1) | 0 (0)
Hypersensitivity (Nervous system disorders) | 1/14 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1/14 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1/14 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1/14 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 1/14 (1) | 0 (0)
Increased appetite (General disorders) | 1/14 (1) | 0 (0)
Influenza like illness (Infections and infestations) | 1/14 (1) | 0 (0)
Inguinal hernia (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 0 (0)
Kidney enlargement (Renal and urinary disorders) | 1/14 (1) | 0 (0)
Libido decreased (Reproductive system and breast disorders) | 1/14 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1/14 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/14 (1) | 0 (0)
Peripheral oedema (General disorders) | 1/14 (1) | 0 (0)
Plantar erythema (Skin and subcutaneous tissue disorders) | 1/14 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1/14 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1/14 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/14 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1/14 (1) | 0 (0)
Syncope (Nervous system disorders) | 1/14 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/14 (1) | 0 (0)
Toothache (General disorders) | 1/14 (1) | 0 (0)
Troponin increased (Cardiac disorders) | 1/14 (1) | 0 (0)
Urine output decreased (Renal and urinary disorders) | 1/14 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0/14 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0/14 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0/14 (0) | 1 (1)
Decreased interest (Nervous system disorders) | 0/14 (0) | 1 (1)
Drooling (Nervous system disorders) | 0/14 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0/14 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0/14 (0) | 1 (1)
Early satiety (Gastrointestinal disorders) | 0/14 (0) | 1 (1)
Eye infection (Infections and infestations) | 0/14 (0) | 1 (1)
Gastroenteritis viral (Gastrointestinal disorders) | 0/14 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0/14 (0) | 1 (1)
Hallucination, auditory (Nervous system disorders) | 0/14 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0/14 (0) | 1 (1)
Hepatic steatosis (Gastrointestinal disorders) | 0/14 (0) | 1 (1)
Hyperhidrosis (Nervous system disorders) | 0/14 (0) | 1 (1)
Infection - Other (DBS lead) (Surgical and medical procedures) | 0/14 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0/14 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0/14 (0) | 1 (1)
Mood altered (Nervous system disorders) | 0/14 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0/14 (0) | 1 (1)
Muscular weakness (General disorders) | 0/14 (0) | 1 (1)
Neurophathy peripheral (Nervous system disorders) | 0/14 (0) | 1 (1)
Nightmare (Nervous system disorders) | 0/14 (0) | 1 (1)
Pernicious anaemia (Blood and lymphatic system disorders) | 0/14 (0) | 1 (1)
Pseudomeningocele (Nervous system disorders) | 0/14 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0/14 (0) | 1 (1)
Pyrexia (Infections and infestations) | 0/14 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0/14 (0) | 1 (1)
Rhinitis allergic (Immune system disorders) | 0/14 (0) | 1 (1)
Sensation of heaviness (Nervous system disorders) | 0/14 (0) | 1 (1)
Sinus congestion (Immune system disorders) | 0/14 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0/14 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/14 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0/14 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0/14 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0/14 (0) | 1 (1)
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 0/14 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0/14 (0) | 1 (1)
Vertigo (Nervous system disorders) | 0/14 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes